CLINICAL TRIAL: NCT06053203
Title: Utilization of Aspirin for Prevention of Pre-Eclampsia in Nigeria: A Explanatory Sequential Mixed Methods Study
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Abuja Teaching Hospital (Other); Aminu Kano Teaching Hospital (Other); Murtala Muhammad Specialist Hospital (Other); National Hospital, Abuja (Other Government)
Responsible Party: Principal Investigator, Zainab Mahmoud, Instructor in Medicine, Division of Cardiology, Washington University School of Medicine
Other Study IDs: NCT-ASPNSTD
Record Dates: First submitted 2023-09-14; First posted 2023-09-25 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-11

CONDITIONS: Hypertensive Disorders of Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- University of Abuja Teaching Hospital: Pregnant women with Hypertensive Disorder of Pregnancy who seek care in the Federal Capital Territory, attending antenatal clinics on the 2nd or subsequent visit and pregnant women presenting to the labor and delivery room.
  Interventions: Other: Exposure of interest - Moderate or High-risk Preeclampsia
- Amino Kano Teaching Hospital: Pregnant women with Hypertensive Disorder of Pregnancy who seek care in Kano State in Nigeria, attending antenatal clinics on the 2nd or subsequent visit and pregnant women presenting to the labor and delivery room.
  Interventions: Other: Exposure of interest - Moderate or High-risk Preeclampsia
- National Hospital, Abuja: Pregnant women with Hypertensive Disorder of Pregnancy who seek care in the Federal Capital Territory, attending antenatal clinics on the 2nd or subsequent visit and pregnant women presenting to the labor and delivery room.
  Interventions: Other: Exposure of interest - Moderate or High-risk Preeclampsia
- Murtala Muhammad Specialist Hospital: Pregnant women with Hypertensive Disorder of Pregnancy who seek care in Kano State in Nigeria, attending antenatal clinics on the 2nd or subsequent visit and pregnant women presenting to the labor and delivery room.
  Interventions: Other: Exposure of interest - Moderate or High-risk Preeclampsia

INTERVENTIONS:
Other: Exposure of interest - Moderate or High-risk Preeclampsia — No intervention

SUMMARY:
The goal of this study is to evaluate the use of aspirin for the prevention of preeclampsia among moderate -to- high-risk pregnant women in tertiary care hospitals in Nigeria followed by a qualitative study to evaluate the barriers and facilitators of aspirin use in prenatal care for the prevention of preeclampsia in Nigeria. The main question[s] it aims to answer are:

1. Is Aspirin used for the prevention of preeclampsia among pregnant women in Nigeria?
2. What factors promote or prevent the utilization of Aspirin for preeclampsia prevention among pregnant women in Nigeria.

DETAILED DESCRIPTION:
Nigeria has the highest burden of maternal mortality worldwide accounting for over 1 in 4 of global maternal deaths. In a 2022 nationwide analysis of maternal outcomes in 76,563 deliveries across referral-level hospitals in Nigeria, hypertensive disorders of pregnancy (HDP) including preeclampsia accounted for 32% of maternal deaths. Studies have linked the pathophysiology of preeclampsia to peripartum cardiomyopathy (PPCM) which is prevalent in Nigeria.5,6 Patients with PPCM were 4 times as likely to have preeclampsia that patients without PPCM. Among known evidence-based interventions for HDP, aspirin prophylaxis stands out as among the most highly effective in preeclampsia prevention. A comprehensive understanding of utilization patterns, or lack thereof, as well as the identification of barriers and facilitators, can inform implementation studies aimed at increasing adoption of this highly effective and cost-effective intervention.

Aims:

1. To conduct a multisite cross-sectional study to evaluate the utilization of aspirin use for the prevention of preeclampsia amongst moderate- to high-risk pregnant women in tertiary care hospitals in Nigeria. We hypothesize that there is underutilization of aspirin for the prevention of preeclampsia amongst pregnant women at moderate- to high-risk of preeclampsia in Nigeria.
2. To conduct a qualitative research study to evaluate facilitators and barriers to aspirin use in prenatal care for prevention of preeclampsia in Nigeria. We hypothesize that there is underutilization of aspirin for the prevention of preeclampsia amongst pregnant women at moderate- to high- risk of preeclampsia in Nigeria.

ELIGIBILITY:
Inclusion Criteria:

* Adult pregnant woman > 18 years old / emancipated pregnant minors (<18years), according to the stipulations of the Nigerian National Health Research Ethics Committee (NRHEC)
* >12 weeks' gestation attending antenatal care clinics on 2nd or subsequent visit
* Those presenting to the labor and delivery room.

Exclusion Criteria:

* Unable to provide consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females who are pregnant
Study Population: Pregnant women attending antenatal clinic or presenting to the labor ward at 2 tertiary and 2 secondary health facilities in the Federal capital territory and Kano state of Nigeria.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Aspirin Use Proportion | 12 weeks- 42 weeks gestation
  Proportion of women (participants) at moderate- or high-risk of preeclampsia who report aspirin use.

SECONDARY OUTCOMES:
Moderate or High-risk Preeclampsia Proportion. | Throughout study duration, from 2nd antenatal visit or after 12 weeks' gestation
  Proportion of women at moderate- to high-risk of preeclampsia among those attending antenatal care who are participants.

OTHER OUTCOMES:
Preeclampsia or Eclampsia proportion categorized as moderate or high risk | Throughout study duration, from 2nd antenatal visit or after 12 weeks' gestation
  Proportion of women presenting with preeclampsia or eclampsia at delivery who would have been categorized as moderate or high- risk at antenatal care visits out of the entire cohort of pregnant participants.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Huffman, MD MPH, Principal Investigator — Washington University School of Medicine; Dike Ojji, MBBS PhD, Principal Investigator — University of Abuja Teaching Hospital; Kathryn Lindley, Principal Investigator — Vanderbilt University
Locations (4):
- Nigeria (4):
  - National Hospital, Abuja, Abuja
  - University of Abuja Teaching Hospital, Gwagwalada
  - Aminu Kano Teaching Hospital, Kano
  - Murtala Muhammad Specialist Hospital, Kano

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available within 1 year of study completion.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 1 year of study conclusion
Access Criteria: After completion of this study, to ensure that our results are used by researchers, policymakers, and community-based organizations, we will disseminate our results through the following:
  * Organize community fora to share results with patients that participated in the study
  * Peer-review all published products with the research team and study partners
  * Report the results at conferences that target researchers, community health providers, and policymakers